CLINICAL TRIAL: NCT00976469
Title: An Open-Label Phase 1/2 Study to Assess the Immunogenicity and Safety of Two Different Dose Levels of H1N1 Pandemic Influenza Vaccine in Healthy Infants, Children and Adolescents Aged 6 Months to 17 Years
Brief Title: A/H1N1 Immunogenicity and Safety in Infants, Children and Adolescents
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alachua Government Services, Inc. (Industry)
Responsible Party: Eva Maria Poellabauer, MD; Study Medical Director, Baxter Healthcare Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 820903; EUDRACT Number 2009-013131-38
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2011-05

CONDITIONS: Influenza; Pandemic Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Licensure; Inflexal V

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dose A (3.75 µg HA antigen, 0.25 mL) (Experimental): Within each age stratum (4 age strata) subjects will be randomized 1:1 to receive two vaccinations of either Dose A (3.75 µg) or Dose B (7.5 µg) of H1N1 pandemic influenza vaccine at a 21-day interval.
  Interventions: Biological: H1N1 pandemic influenza vaccine (whole virion, Vero cell-derived, inactivated)
- Dose B (7.5µg HA antigen, 0.5 mL) (Experimental): Within each age stratum (4 age strata) subjects will be randomized 1:1 to receive two vaccinations of either Dose A (3.75 µg) or Dose B (7.5µg) of H1N1 pandemic influenza vaccine at a 21-day interval. A booster vaccination with a licensed seasonal trivalent influenza vaccine for the season 2010/2011 will be administered to at least 30 subjects in each age stratum (who have received Dose B) at 360 days after the first vaccination.
  Interventions: Biological: H1N1 pandemic influenza vaccine (whole virion, Vero cell-derived, inactivated); Biological: Seasonal trivalent influenza vaccine (licensed) for the season 2010/2011

INTERVENTIONS:
Biological: H1N1 pandemic influenza vaccine (whole virion, Vero cell-derived, inactivated) — 2-dose priming at a 21-day interval, intramuscular injection in either the upper arm or thigh, depending on the subject´s age
Biological: Seasonal trivalent influenza vaccine (licensed) for the season 2010/2011 — Booster vaccination at Day 360 after first vaccination (only in subjects who received the 7.5 µg dose of the H1N1 pandemic influenza vaccine)
  Other Names: Inflexal V
  Arms: Dose B (7.5µg HA antigen, 0.5 mL)

SUMMARY:
The purpose of this study is to determine the preferred dose of H1N1 pandemic influenza vaccine in a pediatric population, aged 6 months to 17 years, based upon assessments of immunogenicity and safety.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided by subject's parent(s) / legal guardian(s) (according to national law)
* Written assent provided by subject according to age and capacity of understanding
* Subject is 9 to 17 years (Stratum A), 3 to 8 years (Stratum B), 12 to 35 months (Stratum C) or 6 to 11 months of age (Stratum D) at the time of screening
* Subject was born at full term of pregnancy (>= 37 weeks) with a birth weight >= 2 kg (Strata C and D) Subject / parent(s) / legal guardian(s) understand(s) the nature of the study and is / are willing to comply with the requirements of the protocol (e.g. return for follow-up visits, completion of the subject diary)
* If female of childbearing potential, subject presents with a negative urine pregnancy test within 24 hours prior to the first vaccination and agrees to employ adequate birth control measures for the duration of the study
* Subject is generally healthy, as determined by the investigator's clinical judgment through collection of medical history and the performance of a physical examination
* Subject is physically and mentally capable of participating in the study

Exclusion Criteria:

* Subject has participated in another clinical study involving an investigational drug, biological product or device within 30 days prior to study enrollment or is scheduled to participate in another clinical study involving an investigational drug, biological product or device during the course of this study
* Subject has a history of exposure to A/H1N1/California/07/2009 virus or a history of vaccination with A/H1N1/California/07/2009 antigen or a closely related influenza virus antigen
* Subject has any inherited or acquired immune deficiency
* Subject currently has or has a recent history of significant neurological, cardiovascular or pulmonary (including asthma), hepatic, metabolic, rheumatic, autoimmune, hematological or renal disorder
* Subject has a history of testing positive for Human Immunodeficiency Virus (HIV), Hepatitis B Surface Antigen (HBsAg) or Hepatitis C Virus (HCV). No confirmatory testing for previous infection with these viruses will be conducted as part of this clinical study.
* Subject has a disease or is currently undergoing a form of treatment or was undergoing a form of treatment within 30 days prior to study entry that could be expected to influence immune response. Such treatment includes, but is not limited to systemic or high dose inhaled corticosteroids, radiation treatment, or other immunosuppressive or cytotoxic drugs.
* Subject has a history of severe allergic reactions or anaphylaxis
* Subject has a rash, dermatologic condition or tattoos which might interfere with injection site reaction rating
* Subject has received a blood transfusion or immunoglobulins within 90 days of study entry
* Subject has received any live vaccine within 4 weeks or inactivated vaccine within 2 weeks prior to vaccination in this study Subject has functional or surgical asplenia
* Subject has a known or suspected problem with alcohol or drug abuse
* Subject or one of subject's parent(s) / legal guardian(s) is in a dependent relationship with one of the study team members. Dependent relationships include close relatives (i.e., children, siblings, partner/spouse, parents) as well as employees of the investigator or site personnel conducting the study
* Subject is pregnant or lactating

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-04 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
To assess the immune response to two different dose levels of a H1N1 pandemic influenza vaccine in healthy infants, children and adolescents aged 6 months to 17 years | 42 days
To assess the safety of two different dose levels of a H1N1 pandemic influenza vaccine in healthy infants, children and adolescents aged 6 months to 17 years | Within 7 days after each vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Eva-Maria Pöllabauer, MD, Study Director — Baxter Healthcare Corporation
Locations (6):
- Austria (3):
  - General Practice, Eferding, Upper Austria
  - General Practice, Wels, Upper Austria
  - Allgemeines Krankenhaus (AKH) der Stadt Wien (General Hospital Vienna), Vienna
- Germany (3):
  - General Practice, Ettenheim
  - General Practice, Kehl
  - General Practice, Mönchengladbach

REFERENCES:
- [Derived] Loew-Baselli A, Pavlova BG, Fritsch S, Poellabauer EM, Draxler W, Kistner O, Behre U, Angermayr R, Neugebauer J, Kirsten K, Forster-Waldl E, Koellges R, Ehrlich HJ, Barrett PN. A non-adjuvanted whole-virus H1N1 pandemic vaccine is well tolerated and highly immunogenic in children and adolescents and induces substantial immunological memory. Vaccine. 2012 Sep 7;30(41):5956-66. doi: 10.1016/j.vaccine.2012.07.039. Epub 2012 Jul 28. PMID 22846396